CLINICAL TRIAL: NCT05084716
Title: PrEP Provision for Ugandan Fisherfolk
Brief Title: Pre-Exposure Prophylaxis (PrEP) Provision for Ugandan Fisherfolk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: Mildmay Uganda Limited (Other); Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R34MH119924 (NIH)
Record Dates: First submitted 2021-10-06; First posted 2021-10-20 (Actual); Results first posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-07

CONDITIONS: HIV
Keywords: PrEP; Fisherfolk; Uganda; HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention (Experimental): At the intervention site during healthcare facility outreach events, all community members will be offered the opportunity to attend intervention workshops where they can learn basic facts about PrEP and be taught skills about how to advocate for PrEP in their community. Check-in reminder calls will be conducted systematically with PrEP users. Healthcare facility staff will encourage PrEP initiators to select an adherence supporter.
  Interventions: Behavioral: Enhanced PrEP provision
- Pre-Intervention Standard of Care (No Intervention): Prior to the intervention period in the intervention community, healthcare facility staff will provide PrEP through outreach events and in local healthcare facilities according to the standard of care.
- Comparison Community (No Intervention): The comparison community will receive standard of care for PrEP provision.

INTERVENTIONS:
Behavioral: Enhanced PrEP provision — At the intervention site during healthcare facility outreach events, all community members will be offered the opportunity to attend intervention workshops where they can learn basic facts about PrEP and be taught skills about how to advocate for PrEP in their community. Check-in reminder calls will be conducted systematically with PrEP users. Healthcare facility staff will encourage PrEP initiators to select an adherence supporter.
  Arms: Intervention

SUMMARY:
This study is a pilot test of enhancements to the standard of care for providing PrEP in Ugandan fishing communities. The specific aims are to conduct a mixed-methods study assessing enhancements to the standard of care for providing PrEP in fisherfolk communities in Lake Victoria, Uganda.

DETAILED DESCRIPTION:
The study will take place at two landing sites at which PrEP is provided to fisherfolk through the Ugandan national PrEP program. The comparison site will receive the standard of care for PrEP provision. At the intervention site, the investigators will implement a three-pronged intervention:

1. During healthcare outreach events we will conduct PrEP workshops, in which people who want to know more about PrEP learn basic facts about PrEP and are taught skills about how to advocate for PrEP in their community.
2. Check-in Calls: To support PrEP adherence, healthcare workers will call PrEP users two weeks after initiation, and the week before refill events, to check in about any questions and to remind them of the next date and place to pick up refills. Calls after PrEP initiation will ask about side effects.
3. To support PrEP adherence, healthcare workers will encourage PrEP users to select an adherence supporter, who is a family member or friend to whom they disclose their PrEP use. The adherence supporter agrees to remind the PrEP user to adhere to PrEP and get refills. Healthcare workers will ask the PrEP user for the name and contact information for the adherence supporter, so that the adherence supporter can be contacted to remind them about refills, as well as if the PrEP user does not show up for a refill.

ELIGIBILITY:
Inclusion Criteria for PrEP initiation:

* Tests HIV-negative at a healthcare outreach/HIV testing event in one of the two selected fishing communities and is PrEP-eligible

Exclusion Criteria:

* Not meeting the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 885 (Actual)
Dates: Start 2021-09-24 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura M Bogart, PhD, Principal Investigator — RAND; Rhoda K Wanyenze, MBChB,PhD,MPH, Principal Investigator — Makerere University
Locations (2):
- Uganda (2):
  - Makerere University School of Public Health, Kampala
  - Mildmay Uganda, Kampala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bogart LM, Musoke W, Mukama CS, Allupo S, Klein DJ, Sejjemba A, Mwima S, Kadama H, Mulebeke R, Pandey R, Wagner Z, Mukasa B, Wanyenze RK. Enhanced Oral Pre-exposure Prophylaxis (PrEP) Implementation for Ugandan Fisherfolk: Pilot Intervention Outcomes. AIDS Behav. 2024 Oct;28(10):3512-3524. doi: 10.1007/s10461-024-04432-w. Epub 2024 Jul 19. PMID 39028385

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at two mainland fisherfolk landing sites in Wakiso District, Uganda. We collected healthcare facility data on HIV testing and PrEP eligibility 6-months before and during the intervention (4-9/21 & 9/21-2/22, respectively) in the intervention community, and during the intervention in the comparison community; and medical records for de-identified client-level PrEP initiation and refill dates for all PrEP users who initiated before and during the intervention (4/21-8/22).
Units Other Than Participants: Community
Groups:
- Intervention Period, Intervention Site: At the intervention site during healthcare facility outreach events, all community members were offered the opportunity to attend intervention workshops where they learned basic facts about PrEP and were taught skills about how to advocate for PrEP in their community. Check-in reminder calls were conducted systematically with PrEP users. Healthcare facility staff encouraged PrEP initiators to select an adherence supporter.
- Pre-intervention Period, Intervention Site: Prior to the intervention period in the intervention community, healthcare facility staff provided PrEP through outreach events and in local healthcare facilities according to the standard of care.
- Intervention Period, Comparison Site: During the intervention period in the comparison community, healthcare facility staff provided PrEP through outreach events and in local healthcare facilities according to the standard of care.
Period: Overall Study
Arm/Group | Intervention Period, Intervention Site | Pre-intervention Period, Intervention Site | Intervention Period, Comparison Site
Started | 199; 1 Community (Note that the pre-intervention participants in the intervention community are different people than the during-intervention participants in the intervention community.) | 142; 1 Community | 544; 1 Community
Completed | 199; 1 Community | 142; 1 Community | 544; 1 Community
Not Completed | 0; 0 Community | 0; 0 Community | 0; 0 Community

BASELINE CHARACTERISTICS:
Groups:
- Intervention Period, Intervention Site: At the intervention site during healthcare facility outreach events, PrEP initiators will be offered guidance on selecting an adherence supporter during PrEP initiation. All outreach event attendees at the events will be offered the opportunity to attend the intervention workshops. Check-in reminder calls will be conducted systematically with PrEP users.
  Enhanced PrEP provision: The intervention will train health care providers to facilitate workshops at outreach events where attendees can learn basic facts about PrEP and be taught skills about how to advocate for PrEP in their community. Healthcare facility staff will encourage PrEP initiators to select an adherence supporter. Check-in reminder calls will be conducted systematically with PrEP users.
- Pre-intervention Period, Intervention Site: Prior to the intervention period in the intervention community, healthcare facility staff will provide PrEP through outreach events and in local healthcare facilities according to the standard of care.
- Intervention Period, Comparison Site: At the control site, healthcare facility staff will continue to provide PrEP according to the standard of care.
- Total: Total of all reporting groups
Arm/Group | Intervention Period, Intervention Site | Pre-intervention Period, Intervention Site | Intervention Period, Comparison Site | Total
Number analyzed (Participants) | 199 | 142 | 544 | 885
Age, Continuous [Mean (Standard Deviation); unit: years] — Age data were obtained from medical records for PrEP users Population: We only had IRB approval to collect demographic data for those who initiated PrEP
  years
    number analyzed (Participants) | 192 | 120 | 426 | 738
    (all) | 31.2 (9.5) | 29.1 (7.9) | 27.3 (5.3) | 28.6 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: We only had IRB approval to collect demographic data for those who initiated PrEP
  Participants
    number analyzed (Participants) | 192 | 120 | 426 | 738
    Female | 105 | 49 | 160 | 314
    Male | 87 | 71 | 266 | 424
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black African | 199 | 142 | 544 | 885

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With PrEP Initiation
Description: Individuals who are eligible for PrEP (tested HIV-negative, aged 18 and older, in fisherfolk community) are asked by a healthcare provider whether they want to start taking PrEP
Time Frame: Baseline. Individuals are asked if they wish to initiate PrEP after they have been tested and deemed eligible
Population: All individuals eligible for PrEP are given the option of initiating (1) or declining (0).
Measure: Count of Participants; unit: Participants
Groups:
- Intervention Period, Intervention Site: At the intervention site during healthcare facility outreach events, all community members will be offered the opportunity to attend intervention workshops where they can learn basic facts about PrEP and be taught skills about how to advocate for PrEP in their community. Check-in reminder calls will be conducted systematically with PrEP users. Healthcare facility staff will encourage PrEP initiators to select an adherence supporter.
- Pre-Intervention Period, Intervention Site: Prior to the intervention period in the same community, healthcare facility staff will provide PrEP through outreach events and in local healthcare facilities according to the standard of care.
- Intervention Period, Comparison Site: During the intervention period in the control community, healthcare facility staff will provide PrEP through outreach events and in local healthcare facilities according to the standard of care.
Arm/Group | Intervention Period, Intervention Site | Pre-Intervention Period, Intervention Site | Intervention Period, Comparison Site
Number analyzed (Participants) | 199 | 142 | 544
Participants | 192 | 120 | 426
Statistical Analysis 1: Comparison: Intervention Period, Intervention Site vs Pre-Intervention Period, Intervention Site; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 5.03, 95% CI 2-sided [2.08 to 12.13]
Statistical Analysis 2: Comparison: Intervention Period, Intervention Site vs Intervention Period, Comparison Site; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 7.60, 95% CI 2-sided [3.48 to 16.59]

2. Primary Outcome: Number of Participants Who Persisted On PrEP After Initiation
Description: Percentage of PrEP users who are still on PrEP at 6 months post-initiation
Time Frame: 6 months
Population: Analysis of PrEP persistence is restricted to those who initiated PrEP
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Period, Intervention Site | Pre-Intervention Period, Intervention Site | Intervention Period, Comparison Site
Number analyzed (Participants) | 192 | 120 | 426
Participants | 92 | 8 | 145
Statistical Analysis 1: Comparison: Intervention Period, Intervention Site vs Pre-Intervention Period, Intervention Site; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 12.88, 95% CI 2-sided [5.96 to 27.85]
Statistical Analysis 2: Comparison: Intervention Period, Intervention Site vs Intervention Period, Comparison Site; Test type: Superiority; p = .001, Regression, Logistic; Odds Ratio (OR) = 1.78, 95% CI 2-sided [1.26 to 2.52]

3. Secondary Outcome: Number of Participants Who Maintained PrEP Prescriptions Over 6 Months
Description: Percentage of PrEP users with a PrEP medication possession ratio of at least 80% coverage by PrEP prescriptions over 6 months. (i.e., 144 of 180 days)
Time Frame: 6 months
Population: Analysis of PrEP coverage is restricted to those who initiated PrEP
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Period, Intervention Site | Pre-Intervention Period, Intervention Site | Intervention Period, Comparison Site
Number analyzed (Participants) | 192 | 120 | 426
Participants | 69 | 0 | 300
Statistical Analysis 1: Comparison: Intervention Period, Intervention Site vs Pre-Intervention Period, Intervention Site; Test type: Superiority; p < .0001, Fisher Exact — Odds Ratio is undefined and p-value from Fisher's Exact test is reported because 0% of PrEP users had ≥80% medication coverage pre-intervention; Cohen's d for difference in proportions = 1.28
Statistical Analysis 2: Comparison: Intervention Period, Intervention Site vs Intervention Period, Comparison Site; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 0.24, 95% CI 2-sided [0.16 to 0.34]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Intervention Period, Intervention Site | Pre-Intervention Period, Intervention Site | Intervention Period, Comparison Site
All-Cause Mortality (participants affected / at risk) | 0/192 | 0/120 | 0/426
Serious Adverse Events (participants affected / at risk) | 0/192 | 0/120 | 0/426
Other Adverse Events (participants affected / at risk) | 0/192 | 0/120 | 0/426

LIMITATIONS AND CAVEATS:
The intervention and comparison communities were mismatched: the comparison community had a less mobile population and a healthcare center (and the intervention community did not), making refill access easier. In addition, pre-intervention PrEP refill data were not available for the comparison site. Thus, we present results for the pre vs. during intervention period comparison in the intervention community, and for the intervention vs. comparison communities during the intervention period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-08): https://cdn.clinicaltrials.gov/large-docs/16/NCT05084716/Prot_SAP_001.pdf
  • Informed Consent Form (2021-07-30): https://cdn.clinicaltrials.gov/large-docs/16/NCT05084716/ICF_002.pdf